CLINICAL TRIAL: NCT06928818
Title: Prospective Observational Study of Trastuzumab Emtansine Immediately After Trastuzumab Deruxtecan in Patients With Advanced Human Epidermal Growth Factor Receptor 2-Positive Breast Cancer in Korea
Brief Title: Trastuzumab Emtansine(T-DM1) After Trastuzumab Deruxtecan(T-DXd) in HER2-Positive Breast Cancer in Korea
Status: Recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Kyung-Hun Lee, Principal Investigator, Seoul National University Hospital
Other Study IDs: H-2412-069-1597
Record Dates: First submitted 2025-03-31; First posted 2025-04-15 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-03

CONDITIONS: Cancer of Breast; Trastuzumab Emtansine; Trastuzumab Deruxtecan
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Prospective observational study of trastuzumab emtansine immediately after trastuzumab deruxtecan in patients with advanced HER2-positive breast cancer in Korea

ELIGIBILITY:
Inclusion Criteria:

* HER2-positive, advanced (unresectable locally advanced or metastatic) breast cancer
* Prior treatment with trastuzumab deruxtecan(T-DXd) in the advanced setting
* Intention to treat with Trastuzumab Emtansine (T-DM1) as first therapy upon T-DXd progression

Exclusion Criteria:

* Any systemic treatment, other than T-DM1, for breast cancer after trastuzumab deruxtecan (As an exception, patients treated with endocrine agents, not in combination with cytotoxics or antibody-drug conjugates, will be permitted in the study)
* Has been previously treated with T-DM1 for advanced breast cancer
* Has been previously treated with 4 or more lines of therapy for advanced breast cancer

  * Half (50%) or more patients will be those who were treated with second-line trastuzumab deruxtecan (i.e. patients at the later line will be capped).

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * Signed Informed Consent Form, when the patient is alive and not lost to follow- up.
  * Age ≥ 19 years old.
  * Histologically or cytologically confirmed, HER2-positive advanced breast cancer which is either locally advanced precluding resection or metastatic.
  * Prior treatment with T-Dxd in the advanced setting
  * Intention to treat with T-DM1 as next therapy upon progression from T-Dxd
  Patients who meet any of the following criteria will be excluded from study entry:
  * Any systemic treatment, other than T-DM1, for breast cancer after T-Dxd (With an exception, endocrine agents not in combination with cytotoxics or antibody-drug conjugates will be permitted in the study)
  * Has been previously treated with T-DM1 for advanced breast cancer
  * Has been previously treated with 4 or more lines of therapy for advanced breast cancer
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | PFS is defined as the time from treatment initiation to the first occurrence of disease progression or death from any cause, whichever occurs first, assessed up to 12 months.
  PFS will be assessed by physicians as per routine clinical practice. CT and/or MRI scans will be at baseline and every 2-4 cycles at the treating physician's discretion, reflecting the observational study design.

SECONDARY OUTCOMES:
objective response rate (ORR) | 12-month
  • objective response rate (ORR)
12-month survival rate | 12-month
  12-month survival rate
time-to-discontinuation (TTD) | 12-month
  time-to-discontinuation (TTD)
time-to-next-line-treatment (TTNT) | 12-month
  time-to-next-line-treatment (TTNT), disregarding endocrine treatments as the maintenance
Duration of therapy (DoT) | 12-month
  Duration of therapy (of T-DM1) will be compared to the duration of previous therapy (T-DXd) to ensure the comparability of each treatments reflecting the tumor biology and clinical course.
Incidence of Treatment-Emergent Adverse Events | 12-month
  Incidence of Treatment-Emergent Adverse Events

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Hospital, Seoul, South Korea